CLINICAL TRIAL: NCT00683332
Title: A Prospective, Observational Study To Monitor Safety In Patients Who Were Administered With Tigecycline (Tygacil) 50 mg By Intravenous Injection (An Observational Study for Safety - Monitored Release)
Brief Title: Post-Marketing Study Of The Safety Of Tygacil (Tigecycline)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Other Study IDs: 3074A1-102235; B1811057
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2011-07-08 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-06

CONDITIONS: Complicated Skin and Skin Structure Infections; Complicated Intra-abdominal Infections
Keywords: Observational study; Tigecycline; infection; skin; abdominal
MeSH Terms: conditions — Infections | interventions — Tigecycline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: Tigecycline (Tygacil)

INTERVENTIONS:
Drug: Tigecycline (Tygacil) — This is a non-interventional study; patients are administered Tygacil as prescribed by their doctor as per registered indications stated in product label/insert (50 mg by Intravenous Injection).

SUMMARY:
The purpose of this study is to collect post-marketing information on the safety of Tygacil in Filipino patients.

DETAILED DESCRIPTION:
Three-thousand or 10% of total number of patients given tigecycline will be included in the study

ELIGIBILITY:
Inclusion Criteria:

* All patients from the study center who received or will receive at least one dose of Tygacil according to the approved product indication.

Exclusion Criteria:

* Previously discontinued Tygacil therapy due to significant safety concern.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who receive one dose of tigecycline
Sampling Method: Non-Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2007-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Manila, Philippines

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3074A1-102235&StudyName=Post-Marketing%20Study%20Of%20The%20Safety%20Of%20Tygacil%20%28Tigecycline%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Tygacil 50 mg: Filipino participants received at least 1 intravenous (IV) dose of tygacil 50 mg administered per registered indication as stated in the product label/insert
Period: Overall Study
Arm/Group | Tygacil 50 mg
Started | 621
Completed | 621
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tygacil 50 mg
Number analyzed (Participants) | 621
Age Continuous [Mean (Standard Deviation); unit: Years] | 55.7 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254
  Male | 367

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Spontaneous Adverse Events
Description: Adverse events were based on the signs or symptoms detected during the physical examination and on clinical evaluation of the participant. In addition to the information obtained from these sources, the participant was asked the following nonspecific question: "How have you been feeling since your last visit?"
Time Frame: 30 days post injection up to 3 years
Population: Safety Population: All participants who received at least 1 dose of tygacil
Measure: Number; unit: Participants
Arm/Group | Tygacil 50 mg
Number analyzed (Participants) | 621
Participants | 17

ADVERSE EVENTS:
Time Frame: 30 days post injection up to 3 years
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Tygacil 50 mg
Serious Adverse Events (participants affected / at risk) | 5/621
Other Adverse Events (participants affected / at risk) | 12/621
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tygacil 50 mg (N=621)
Cardiopulmonary Arrest (Cardiac disorders) | 4
Haematuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tygacil 50 mg (N=621)
Eosinophilia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Phlebitis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.